CLINICAL TRIAL: NCT06411418
Title: Evaluation of Flow Diverter Technology Device for Intracranial Aneurysm
Acronym: SHIELD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: Jacobs institute (Other)
Responsible Party: Principal Investigator, Elad Levy, Principal Investigator, State University of New York at Buffalo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Version 2.0
Record Dates: First submitted 2024-04-15; First posted 2024-05-13 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-10

CONDITIONS: Intracranial Aneurysms
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single arm study (Experimental): Occurrence of thromboembolic event(s)
  Interventions: Device: Pipeline™ Flex Embolization Device with Shield Technology™

INTERVENTIONS:
Device: Pipeline™ Flex Embolization Device with Shield Technology™ — The Pipeline™ Flex Embolization Device with Shield Technology™ for the endovascular treatment of adults (22 years of age or older) with large or giant wide-necked intracranial aneurysms (IAs) in the internal carotid artery from the petrous to the superior hypophyseal segments. The Pipeline™ Flex Embolization Device with Shield Technology™ is also indicated for use in the internal carotid artery up to the terminus for the endovascular treatment of adults (22 years of age or older) with small and medium wide-necked (neck width ≥ 4 mm or dome-to-neck ratio < 2) saccular or fusiform intracranial aneurysm (IAs) arising from a parent vessel with a diameter ≥ 2.0 mm and ≤ 5.0 mm.

SUMMARY:
The Jacobs Institute is participating in a study designed to collect prospective clinical evidence to evaluate the approved use of the Pipeline™ Flex Embolization Device with Shield Technology™ for the endovascular treatment of adults (22 years of age or older) with wide-necked intracranial aneurysms

DETAILED DESCRIPTION:
The Pipeline™ Flex Embolization Device with Shield Technology™ for the endovascular treatment of adults (22 years of age or older) with large or giant wide-necked intracranial aneurysms (IAs) in the internal carotid artery from the petrous to the superior hypophyseal segments. The Pipeline™ Flex Embolization Device with Shield Technology™ is also indicated for use in the internal carotid artery up to the terminus for the endovascular treatment of adults (22 years of age or older) with small and medium wide-necked (neck width ≥ 4 mm or dome-to-neck ratio < 2) saccular or fusiform intracranial aneurysm (IAs) arising from a parent vessel with a diameter ≥ 2.0 mm and ≤ 5.0 mm.

ELIGIBILITY:
Inclusion Criteria:

* Adults (22 years of age or older) with large or giant wide-necked intracranial aneurysms (IAs) in the internal carotid artery from the petrous to the superior hypophyseal segments.

Exclusion Criteria:

* Cannot provide consent or legally authorized representative not available to provide consent

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Occurrence of thromboembolic event(s) | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Elad LEvy, MD, Principal Investigator — University at Buffalo Neurosurgery
Locations (1):
- University at Buffalo Neurosurgery, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No